CLINICAL TRIAL: NCT03088124
Title: Active Surveillance With or Without a 6 Months Apalutamide Treatment in Low Risk Prostate Cancer: A Phase II Randomized Multicenter Trial
Brief Title: Active Surveillance With or Without Apalutamide Treatment in Low Risk Prostate Cancer
Acronym: PC-ARN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC-ARN IPC-2015-025
Record Dates: First submitted 2017-03-13; First posted 2017-03-23 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Low Risk Prostate Cancer
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active surveillance (No Intervention): Active surveillance without androgen deprivation
- active surveillance with Apalutamide (Experimental): Active surveillance during and after 6 months treatment with Apalutamide
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — Patients will take orally everyday 240 mg of Apalutamide.
  Other Names: ARN-509
  Arms: active surveillance with Apalutamide

SUMMARY:
Many prostate cancer are slow or non progressive forms that would never impair quality or quantity of like of life if undetected. For this localized prostate cancer, the recommendation is an active surveillance, however often experienced by the patient as a lack of care. Thus the introduction of new potent androgen receptor inhibitor raise the question of the benefit of early hormonal therapy in localized prostate cancers.

The aim of this study is to assess whether treatment with an oral androgen receptor inhibitor could influence the progression of localized prostate cancer and delay the time to local treatment initiation.

DETAILED DESCRIPTION:
Several cohort studies have demonstrated that survival time in patients with untreated early stage prostate cancer is greater than 10 years in more than 70% of cases, suggesting the existence of slowly progressive or non-progressive forms of prostate cancer that would never cause any impairment to quality or quantity of life if undetected. These forms represent currently 23% to 67% of all prostate cancers. Therefore, while men's lifetime risk of prostate cancer is high (16-18%), the corresponding risk of death is only about 3%. These observations gave the opportunity to consider, near the current standard and curative treatment, an active surveillance. This therapeutically choice offers the ability to delay or avoid definitive treatment, thereby minimizing patient morbidity. Studies to date have shown that this seems to be achieved without compromising long term outcomes (progression-free survival) in appropriately selected patients. Up to one third of them receive further treatment after a median of about 2,5 years of surveillance. However, even if active surveillance is associated with the highest quality-adjusted life expectancy when compared with local treatment, active surveillance is often experienced as a lack of care, some patients undergoing surveillance experience disutility related to anxiety which can significantly affect their quality of life.

The introduction of new potent androgen receptor inhibitors able to block several steps in the androgen receptors signaling pathway, raise the question again of the benefit of early hormonal therapy in localized prostate cancers. The aim of this study is to assess whether treatment with an oral androgen receptor inhibitor could influence the progression of localized prostate cancer and delay the time to local treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Out-patient aged ≥ 18 years old
2. With life expectancy of more than 5 years
3. With ECOG performance status = 0 or 1
4. Having read, understood, signed and dated the informed consent,
5. With a Localized prostate cancer diagnozes within less than 7 months and defined by:

   * Clinical Stage: T1c or T2a
   * Sampled biopsy with less of 3 positive cores and tumor length < 3 mm per core (<7 mm for targeted cores)
   * Gleason score < 7 (3+4 for patients >70years if small volume tumor)
   * PSA levels ≤ 10 ng/ml or PSA density <0.2ng/ml/ml
6. Clinical laboratory values at screening:

   1. Hemoglobin ≥9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
   2. Platelet count ≥100,000 x 109/µL independent of transfusion and/or growth factors within 3 months prior to randomization
   3. Serum albumin ≥3.0 g/dL
   4. Serum creatinine <2.0 × upper limit of normal (ULN)
   5. Serum potassium ≥3.5 mmol/L
   6. Serum total bilirubin ≤1.5 × ULN (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject may be eligible)
   7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 × ULN
7. Medications known to lower the seizure threshold (see list in appendix 2) must be discontinued or substituted at least 4 weeks prior to study entry.
8. Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
9. Having accepted the principle of active surveillance
10. Who is willing to participate to the study for a minimum period of 36 months
11. Able to swallow the study drug and comply with study requirements
12. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen.

Exclusion Criteria:

1. Prior treatment for prostate cancer with surgery or radiotherapy or including 5-alpha reductase inhibitor (finasteride or dutasteride) and antiandrogen
2. Absolute neutrophil count < 1,500/μL,
3. Seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
4. Any prior malignancy (other than adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) within 5 years prior to randomization
5. Severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
6. Uncontrolled hypertension (SBP≥160 mmHg or DBP≥90 mmHg). Patients with a history of uncontrolled hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
7. Gastrointestinal disorder affecting absorption
8. Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis) or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
9. Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures
10. Mental deficiency or any other reason that may hinder the understanding or the strict application of the Protocol
11. Patient placed under judicial protection, tutorship, or curatorship
12. Patient unlikely to attend control visits
13. Patient currently enrolled in an investigational study or having participated to another investigational study within the past 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Time to initiate a local treatment. | from randomization to local treatment initiation (up to 3 years)
  Date of randomization and date at which local treatment is initiated

SECONDARY OUTCOMES:
Time to another prostate treatment initiation (excluding local treatment) | from randomization to prostate treatment initiation up to 3 years
  Date of randomization, date of treatment initiation (other than local)
Prostate Specific Antigen (PSA) and Testosterone dosages | PSA: at screening and at 3, 6, 9,12,18, 24, 30, 36 months visits. Testosterone: at screening, 12, 24 and 36 months visits
  Biological assessment
Prostate biopsy and Gleason score | At screening and at 12, 24 and 36 months visits
  histological assessment
Tumor radiological progression | At screening and at 24 months-visit
  Radiological assessment by multi-parametric MRI: normal versus anormal

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle GRAVIS, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (11):
- France (11):
  - Institut Paoli Calmettes, Marseille, Bouches Du Rhône
  - CHRU Hopital Edouard Herriot, Lyon
  - Clinique Beau Soleil, Montpellier
  - Chu Hotel Dieu, Nantes
  - Chu de Nice, Nice
  - Institut Mutualiste Montsouris, Paris
  - Chu Tenon, Paris
  - Clinique La Croix Du Sud, Quint-Fonsegrives
  - Chu Pontchaillou, Rennes
  - Chu Saint Etienne, Saint-Etienne
  - Hia Sainte Anne, Toulon

REFERENCES:
- See also: Official web site of the sponsor — http://institutpaolicalmettes.fr